CLINICAL TRIAL: NCT04723095
Title: Establishing a Tumor Registry for Patients With Neuroendocrine Carcinoma of the Cervix
Acronym: NeCTuR
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA12-1006; NCI-2020-07408 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA12-1006 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-13; First posted 2021-01-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cervical Large Cell Neuroendocrine Carcinoma; Cervical Neuroendocrine Carcinoma; Cervical Small Cell Carcinoma; Cervical Undifferentiated Carcinoma; Stage I Cervical Cancer AJCC v8; Stage IA Cervical Cancer AJCC v8; Stage IA1 Cervical Cancer AJCC v8; Stage IA2 Cervical Cancer AJCC v8; Stage IB Cervical Cancer AJCC v8; Stage IB1 Cervical Cancer AJCC v8; Stage IB2 Cervical Cancer AJCC v8; Stage II Cervical Cancer AJCC v8; Stage IIA Cervical Cancer AJCC v8; Stage IIA1 Cervical Cancer AJCC v8; Stage IIA2 Cervical Cancer AJCC v8; Stage IIB Cervical Cancer AJCC v8; Stage III Cervical Cancer AJCC v8; Stage IIIA Cervical Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Chromatin Immunoprecipitation Sequencing; Follow-Up Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical chart review): Patients' medical records are reviewed retrospectively and prospectively. All prospective patients will be contacted via email, telephone, or U.S. Mail on case by case basis for up to 10 years to check status of disease and any further treatment received. Project staff can also access the patient's M. D. Anderson Epic medical record for updates. Request for additional clinic and treatment notes will be submitted to external medical institutions listed in the physician information form in order to access updated notes for non- M. D. Anderson patients.
  Interventions: Other: Follow-Up; Other: Medical Chart Review

INTERVENTIONS:
Other: Follow-Up — Receive follow up
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; Followed; Followup
Other: Medical Chart Review — Review of medical records
  Other Names: Chart Review

SUMMARY:
This study collects information and data on patients with neuroendocrine cervical cancer. Information from this study may be used to better understand the correlation between clinical data, such as patient characteristics, treatment, and disease outcomes, and overall patient outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect, both prospectively and retrospectively, data on disease characterization, treatment, and outcomes for patients with neuroendocrine carcinoma of the uterine cervix.

II. To organize clinical information in order to support multifaceted queries of patient characteristics, treatment, and disease outcome data and to facilitate correlation of these characteristics with patient outcome.

III. To have a single data repository kept on a secure platform that will integrate clinical information and research findings and serve as an archive for future research.

OUTLINE:

Patients' medical records are reviewed retrospectively and prospectively. All prospective patients will be contacted via email, telephone, or U.S. Mail on case by case basis for up to 10 years to check status of disease and any further treatment received. Project staff can also access the patient's M. D. Anderson Epic medical record for updates. Request for additional clinic and treatment notes will be submitted to external medical institutions listed in the physician information form in order to access updated notes for non- M. D. Anderson patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with a personal history of cervical cancer with any portion of neuroendocrine component (including mixed tumors) of the following histologic subtypes:

  * Small cell neuroendocrine carcinoma
  * Large cell neuroendocrine carcinoma
  * Undifferentiated high-grade neuroendocrine carcinoma
* Patients may be in any stage of treatment, surveillance or recurrence at the time of initial participation in the study
* Patients with all stages of disease are considered eligible
* Patients who do not speak English can be eligible if accompanied by an institutional interpreter
* Patients who are receiving or have received treatment at any facility, including but not limited to M. D. Anderson Cancer Center are eligible
* Patient may be residents of any country and be of any ethnic background
* Patients who request to participate in the study, regardless of the method by which they learned of it, are eligible to participate, including, but not limited to patients who seek participation via the website
* Next of kin or legal authorized representatives of patients who are deceased but had a history of neuroendocrine carcinoma (NEC) of the cervix are eligible to participate
* Next of kin or legal authorized representatives of patients must read and speak English

Exclusion Criteria:

* Patients with other histologic subtypes of NEC of the cervix including typical and atypical carcinoid tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with neuroendocrine cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2013-05-16 (Actual); Primary Completion 2044-01-01 (Estimated); Study Completion 2044-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease characterization data | through study completion, an average of 1 year
  Information collected from retrospective and prospective review of medical records.
Patient treatment data | through study completion, an average of 1 year
  Information collected from retrospective and prospective review of medical records.
Patient outcome data | through study completion, an average of 1 year
  Information collected from retrospective and prospective review of medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa A. Meyer, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org